CLINICAL TRIAL: NCT07170787
Title: Phase Ib/II Clinical Study of IMM2510 for Injection Combined With IMM01 for Injection in Advanced Solid Tumors
Brief Title: A Study of IMM2510 + IMM01 Combination Therapy in Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ImmuneOnco Biopharmaceuticals (Shanghai) Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ImmuneOncoBioShanghai
Record Dates: First submitted 2025-09-02; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: Dose Escalation Phase:
  Participants will receive IMM2510 10 mg/kg or 20mg/kg and combine with IMM01 1.0 mg/kg , 2.0 mg/kg or 3.0 mg/kg dose every 2 weeks (Q2W).
  Dose Expansion Phase:
  The dose of IMM2510 and IMM01 for the dose expansion phase is determined according to the dose escalation results.
  Participants will receive IMM2510 and IMM01 every 2 weeks (Q2W).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cohort 1 (Experimental): Dose Escalation Phase:
  Participants will receive IMM2510 10.0 mg/kg or 20.0 mg/kg dose every 2 weeks (Q2W), and will receive IMM01 1.0 mg/kg,2.0 mg/kg or 3.0 mg/kg dose every 2 weeks (Q2W).
  Cohort Expansion Phase:
  The dose of IMM2510 and IMM01 for the cohort expansion phase is determined according to the dose escalation results.
  Participants will receive IMM2510 and IMM01 every 2 weeks (Q2W).
  Interventions: Biological: IMM2510; Biological: IMM01

INTERVENTIONS:
Biological: IMM2510 — IMM2510 administered intravenously once every 2 weeks (Q2W). Dose escalation cohorts will receive ascending doses of IMM2510 (e.g., 10 mg/kg, 20 mg/kg, up to maximum tolerated dose or recommended phase 2 dose).
Biological: IMM01 — IMM01 administered intravenously once every 2 weeks (Q2W). Dose escalation cohorts will receive ascending doses of IMM01 (e.g., 1 mg/kg, 2 mg/kg, 3mg/kg, up to maximum tolerated dose or recommended phase 2 dose).

SUMMARY:
This is a Phase 1, open-label, dose-escalation and cohort expansion study designed to evaluate the safety, tolerability, pharmacokinetics, and preliminary antitumor activity of IMM2510(Anti-PD-L1 and VEGF trap recombinant protein) combine with IMM01(Anti-CD47 Recombinant Protein) in patients with advanced solid tumors who have received at least first line treatment in past.

ELIGIBILITY:
Inclusion Criteria:

* Participant has provided informed consent prior to initiation of any study specific activities/procedures.
* Age greater than or equal to 18 years old at the same time of signing the informed consent.
* Histologically or cytologically confirmed for Solid Tumor.
* Eastern Cooperative Oncology Group (ECOG) 0 to 1.
* Adequate organ function as defined in protocol.

Exclusion Criteria:

* History of other malignancy within the past 5 years with exceptions.
* Systemic chemotherapy was administered within 3 weeks prior to the first administration.
* Activated symptomatic brain metastases and leptomeningeal disease.
* History of inflammatory bowel disease.
* Participants with symptoms and/or clinical signs and/or uncontrolled active systemic infection within 14 days prior to the first dose of study treatment.

Participant has known active infection requiring parenteral antibiotic treatment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2029-02 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
DLT/MTD (Dose Escalation Phase) | Within 28 days after the investigational products administration (within 56 days after first dosing of C1D1)
Incidence and characteristics of AEs and SAEs (according to NCI CTCAE 5.0) | From the first dose to 30 days after the last dose [90 days for SAEs and Immune-related Adverse Event (irAEs) ], or until beginning new anti-tumor treatment
Objective Response Rate (ORR) | From date of first dose until the date of first documented progression, death from any cause, loss of follow-up, withdrawal of informed consent, or study termination by the sponsor, whichever came first, assessed up to approximately 2 years.
RP2D (Dose Extension Phase) | From the first dose until disease progresses or end of treatment for other reasons, the maximum treatment duration is not more than 96 weeks

SECONDARY OUTCOMES:
Disease Control Rate(DCR) | From date of first dose until the date of first documented progression, death from any cause, loss of follow-up, withdrawal of informed consent, or study termination by the sponsor, whichever came first, assessed up to approximately 2 years.
Duration of Response (DOR) | From date of first dose until the date of first documented progression, death from any cause, loss of follow-up, withdrawal of informed consent, or study termination by the sponsor, whichever came first, assessed up to approximately 2 years.
progression- free survival(PFS) | From date of first dose until the date of first documented progression, death from any cause, loss of follow-up, withdrawal of informed consent, or study termination by the sponsor, whichever came first, assessed up to approximately 2 years.
overall survival（OS） | From date of first dose until the date of first documented progression, death from any cause, loss of follow-up, withdrawal of informed consent, or study termination by the sponsor, whichever came first, assessed up to approximately 2 years.
Cmax | Up to approximately 1 year
  Peak concentration (Cmax)
Tmax | Up to approximately 1 year
  Peak time (Tmax)
AUC0-tlast | Up to approximately 1 year
  Area under plasma concentration-time curve from 0 to the last quantifiable time point (AUC0-t)
AUC0-inf | Up to approximately 1 year
  Area under plasma concentration-time curve from 0 to infinite time
t1/2 | Up to approximately 1 year
  Elimination phase half-life (t1/2), in single dose period.
CL | Up to approximately 1 year
  Clearance Rate

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Gobroad Cancer Hospital China Pharmaceutical University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No